CLINICAL TRIAL: NCT03587363
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of Erdafitinib
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of Erdafitinib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Mild/moderate hepatic impairment (HI) cohorts completed with no impact to erdafitinib exposure. Severe HI cohort enrollment stopped early.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108483; 2018-001104-11 (EudraCT Number); 42756493EDI1008 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-07-04; First posted 2018-07-16 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive 6 milligram (mg) erdafitinib as a single oral dose under fasted conditions on Day 1.
  Interventions: Drug: Erdafitinib
- Cohort 2: Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (Child-Pugh score of 5 or 6) will receive 6 mg erdafitinib as a single oral dose under fasted conditions on Day 1.
  Interventions: Drug: Erdafitinib
- Cohort 3: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh score of 7 to 9) will receive 6 mg erdafitinib as a single oral dose under fasted conditions on Day 1.
  Interventions: Drug: Erdafitinib
- Cohort 4: Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment (Child-Pugh score of 10 to 15) will only be enrolled to receive appropriate dose level of erdafitinib after review of preliminary safety and pharmacokinetic (PK) data from the mild and moderate hepatic impairment cohorts.
  Interventions: Drug: Erdafitinib

INTERVENTIONS:
Drug: Erdafitinib — Participants will receive 6 mg (2*3 mg tablet) erdafitinib as a single oral dose on Day 1. Participants in Cohort 4 may receive a lower dose if warranted by preliminary safety and PK data from Cohorts 2 and 3.
  Other Names: JNJ-42756493

SUMMARY:
The primary purpose of the study is to characterize the single dose pharmacokinetic of erdafitinib in participants with impaired hepatic function relative to participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman must have a clinically stable hepatic function as confirmed by the serum bilirubin and transaminase levels measured during screening and those measured on Day -1
* If a woman (a) must not be of childbearing potential postmenopausal or surgically sterile (b) must agree to not donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 3 months after the study drug administration
* If a woman who is considered surgically sterile but not postmenopausal, must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening (exemptions: pregnancy test not required in female participants with prior hysterectomy or prior bilateral oophorectomy)
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 3 months after the study drug administration
* Participants with hepatic impairment must meet the Child-pug classification for mild, moderate or severe hepatic impairment and must have stable hepatic function

Exclusion Criteria:

* History or current evidence of ophthalmic disorder, such as central serous retinopathy (CSR) or retinal vein occlusion, active wet age related macular degeneration, diabetic retinopathy with macular edema, uncontrolled glaucoma, corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration
* Any surgical or medical condition that may alter the absorption, metabolism, or excretion of the study drug (example, gastrectomy, Crohn's disease etc), with the exception of hepatic impairment
* History of drug abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 6 months before screening or positive test result(s) for drugs of abuse (including barbiturates, opiates, cocaine, cannabinoids, amphetamines, hallucinogens, and benzodiazepines) at screening and on Day -1
* Known allergy to the study drug or any of the excipients of the formulation (Physical Description of Study Drug[s], for a list of excipients)
* Donated blood or blood products or had substantial loss of blood (more than 500 milliliter [mL]) within 3 months before study drug administration or intention to donate blood or blood products during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to 21 days
  Cmax is the maximum observed plasma concentration.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) | Up to 21 days
  Tmax is the time to reach maximum observed plasma concentration.
Area Under Plasma Concentration-Time Curve (AUC) | Up to 21 days
  AUC is area under plasma concentration-time curve.
Terminal Elimination Half-life (t1/2term, Lambda) | Up to 21 days
  t1/2term, Lambda is elimination half-life associated with the terminal slope (Lambda[Z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda(Z).
Total Plasma Clearance (CL/F) | Up to 21 days
  CL/F is total plasma clearance of drug after extravascular administration, uncorrected for absolute bioavailability (BA), calculated as Dose/AUC (0-infinity).
Apparent Volume of Distribution (Vd/F) | Up to 21 days
  Vd/F is apparent volume of distribution after extravascular administration, uncorrected for absolute BA.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Approximately 50 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily have a causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel GmbH, Kiel
  - APEX GmbH, München